CLINICAL TRIAL: NCT04725565
Title: Genetics Adviser: Evaluating a Digital Decision Support Tool for Genetic Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3400
Record Dates: First submitted 2021-01-13; First posted 2021-01-26 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: Incidental Findings; Genomic Sequencing; Randomized Controlled Trial; Decision Aid; Clinical Utility; Personal Utility
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genetics ADviSER Decision Aid Plus Standard Genetic Counselling (Experimental): Participants in the intervention arm will use the Genetics ADviSER to learn about genomic sequencing and to select which results they would like to receive from genomics sequencing results. After using the Genetics ADviSER decision aid they will speak with genetic counselor to discuss their choices and to finalized their selection.
  Interventions: Behavioral: Genetics ADvISER Decision Aid Plus Standard Genetic Counselling
- Standard Genetic Counselling Only (Active Comparator): Participants will speak with a genetic counsellor over the phone to learn about genomic sequencing and select which incidental findings they would like to receive from genomic sequencing.
  Interventions: Behavioral: Standard Genetic Counseling

INTERVENTIONS:
Behavioral: Genetics ADvISER Decision Aid Plus Standard Genetic Counselling — The decision aid will educate patients about the types of incidental finding they can learn from genomic sequencing and will give them opportunity select what types of results they would like to receive.
  Arms: Genetics ADviSER Decision Aid Plus Standard Genetic Counselling
Behavioral: Standard Genetic Counseling — Standard Genetic counseling to learn about and select incidental results from genomic sequencing.
  Arms: Standard Genetic Counselling Only

SUMMARY:
Oncologists are increasingly using genomic sequencing to diagnose and optimize care for their patients. A consequence of this technology is its capacity to detect a patient's risk for thousands of current and future conditions or diseases. Guidelines recommend doctors allow patients to choose which results they wish to receive before ordering the test. It is not feasible to counsel patients on the thousands of possible results because of the limited clinical resources and genomics expertise. Decision aids (DAs) can fill this gap, however there are no DAs to guide patients' decisions about results from genomic sequencing. A DA prototype was developed (GenomicsADvISER.com), the first DA of its kind. This study will transform the DA prototype into an interactive, adaptable and patient-centred digital decision support tool (Genetics ADvISER) via user-centred design methods. The objective of this study is to evaluate the effectiveness of Genetics ADvISER in an RCT with patients being offered results from genomic sequencing. Results of this trial will be used to establish whether the Genetics ADvISER is effective to use in practice. This could fill a critical clinical care gap, improve health outcomes and service use by reducing counselling burden as well as overuse, underuse and misuse - concerns of policy makers seeking to address the triple aims of health care.

DETAILED DESCRIPTION:
BACKGROUND: Genomic sequencing (GS) is a driver of precision oncology. Oncologists are increasingly using tumour GS for precision oncology care, which is often times accompanied by germline GS on normal control tissue. One complex feature of this technology is its capacity to generate incidental findings (IF). Guidelines recommend doctors inform patients of their incidental GS results. Yet there are limited tools to communicate the scope and implications of the thousands incidental results available to help guide patients' decisions about which results they wish to learn.

RATIONALE: There are limited decision support tools in genetics. Despite the long-standing practice of medical genetics, there are relatively few decision support tools for genetic testing and very few that have been rigorously evaluated. Even fewer decision support tools exist on possible results from genomic sequencing; existing tools target pediatric contexts, focus on genomic sequencing education-only or on the return of results; they do not cover all possible results with decision support to simulate genetic counselling, limiting their use and applicability in clinical care. Thus, there are no decision support tools to guide patients about all results available from genomic sequencing.

OBJECTIVES: Evaluate the effectiveness of the Genetics ADvISER vs standard genetic counseling (GC) with patients receiving incidental findings.

HYPOTHESIS: Use of the Genetics ADvISER will reduce patients' decisional conflict & anxiety, improve patient knowledge, satisfaction with decisions and preparedness for decision-making when selecting IF compared to GC alone.

PHASE 1: RCT to evaluate the Decision Aid

Methods: This is a mixed method, non-blinded randomized controlled superiority trial. We will evaluate whether use of the Genetics ADvISER followed by Genetic Counsellor (GC) reduces decisional conflict compared to GC alone in a RCT. As a part of this trial, patients will receive results from exome sequencing.

Study population: Adult cancer patients who have had GS for their cancer (but did not receive incidental findings) or adult patients who have had a negative genetic panel test and may eligible for GS.

Sample: The primary outcome is decisional conflict; the study requires 64 patients/arm (128 total) to detect the minimal clinically important difference (MCID) of 0.3 using the Decisional Conflict Scale (DCS), assuming a standard deviation of 0.6, an alpha of 0.05 (two-sided) and power of 0.8. Participants will be consecutively randomized and allocated from an existing list of eligible subjects using a computer-generated randomization in a 1:1 ratio with random permuted blocks of varying sizes. Patients from each clinic will be randomized separately to ensure we have an even distribution of this population in both arms of the study.

Intervention: Participants in the intervention arm will use the Genetics ADviSER to learn about GS, select which results they would like to receive and to receive their GS results.

Control: Participants in the control arm will speak with a genetic counsellor to learn about GS, select which results they would like to receive and to receive their GS results.

Outcomes and measures: The primary outcome is decisional conflict, assessed via the validated Decisional Conflict Scale (DCS) consistent with the ODSF.

Secondary outcomes: Knowledge, measured using an established questionnaire assessing benefits and limitations of genome sequencing and a set of internally developed knowledge questions on IF; Satisfaction with decision-making, measured using the Satisfaction with Decision scale and the Preparation for Decision Making scale; Anxiety, measured using the state subscale of the State-Trait Anxiety Inventory. All sessions will be recorded to assess the length of GC sessions.

Quantitative Analysis: The analysis of outcomes will follow the intention-to-treat approach. Mean scores for decisional conflict, satisfaction with and preparation for decision-making, knowledge of IF and GC session length will be compared using a t-test. Anxiety, knowledge of sequencing benefits and sequencing limitations scores will be assessed by summing the number of correct responses to the questions, and compared adjusting for baseline score using analysis of covariance (ANCOVA). The primary time points of comparison will be (T1) for the control versus (T2) for the intervention group. Secondary exploratory analyses will examine the impact that the decision aid had alone (T1), without the addition of follow-up GC at T2 and at T3, after participants have received their IF on decision conflict, knowledge, anxiety, satisfaction and preparation with decision-making. Descriptive statistics will be used to describe participants' demographic characteristics (age, sex, education, etc.).

PHASE 2: Qualitative study

This study will explore the utility the of the Genetics ADvISER and incidental results via qualitative interviews with participants. After the study is completed, a subset set of participants (n = 40) will be selected to participate qualitative portion of the study. Participants approached to complete the qualitative portion of the study will determined by purposeful sampling, in order to get mix of participants across a range of experiences and demographic characteristics.

Qualitative Analysis: The qualitative analyses will draw on grounded theory. Open coding, constant comparison and axial coding will be used to identify common and divergent themes to characterize the entire dataset. Interviews will consider participants' socio-demographic factors that may influence their informational and decisional needs as well as how they engage with genetic information and participate in shared decision making. Two researchers will code transcripts independently; consensus on codes will be reached through discussion. Validation methods may include triangulation and member checking. In keeping with qualitative methodology, data analysis will occur in conjunction with data collection. On-going analysis will inform the development of progressive iterations of the interview guides.

ELIGIBILITY:
Inclusion Criteria:

* Previous control participants from the Incidental Genomics study who have given permission to be re-contacted for related research or a patient who has undergone germline genetic testing (single gene or panel) and received a negative or inconclusive result.
* 18 years old or older
* Speak and read English.

Exclusion Criteria:

For participants newly recruited (not part of parent trial CTO# 0819)

* Received positive panel testing or panel sequencing
* Have not had germline single gene testing related to their primary cancer condition (e.g., BRCA1/2 for breast/ovarian cancer, MLH, MSH, PMS colorectal cancer, etc.)
* Received a positive germline genetic test for a cancer gene mutation (e.g., BRCA1/2, MLH, MSH, PMS, APC, MUTYH, etc.)
* Currently under cancer treatment
* In stage 4, progressive metastatic cancer

For all

* Do not speak or read English
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Scale (DCS) | 1 day
  The Ottawa Decision Support Framework measure of decisional conflict, a 16 item scale - developed by O'Connor et al. Each item is scored 1-5 and a total score on the DCS is calculated by summing all items on the DCS and then dividing by 16, giving a final score between 1 and 5. A lower score on the DCS indicates lower level of decisional conflict.

SECONDARY OUTCOMES:
Knowledge | Assessed at baseline, immediately after baseline/ post intervention, at two weeks, 2 months and 4 months.
  Knowledge is measured using a genomics knowledge scale developed by Clinseq, an established 11-item questionnaire consisting of two subscales assessing benefits and limitations of genome sequencing. Responses are on a five-point Likert scale ranging from strongly agree to strongly disagree, with responses being assigned a value of 1-5. Higher knowledge score s indicates a higher level of knowledge.
Satisfaction with Decision Scale (SWD) | Assessed immediately after baseline/ post intervention, at two weeks, 2 months and 4 months.
  A six item scale measures a patient satisfaction with a health care decision. Items are scored 1-4. A higher score signifies a higher level of satisfaction or preparation with a decision. Items can be summed and scored (sum the 6 items and divide by 6).
Preparation for Decision Making scale (PrepDM) | Assessed immediately after baseline/ post intervention, at two weeks, 2 months and 4 months.
  A 10 item scale assesses a patient's perception of how useful a decision aid or other decision support intervention is in preparing the respondent to communicate with their practitioner at a consultation visit and making a health decision. Items are scored 1-4. Items can be summed and scored (sum the 10 items and divide by 10). A higher score indicates a higher level of preparation.
State-Trait Anxiety Inventory | Assessed at baseline, immediately after baseline/ post intervention, at two weeks, 2 months and 4 months.
  Measured using the 20 item State-trait scale. Anxiety was measured using the state subscale of the State-Trait Anxiety Inventory. Items can be summed and scored (sum the 20 items and divide by 20). Higher scores on the State-Trait Anxiety Inventory indicate higher level of anxiety.
Hospital Anxiety and Depression Scale (HADS) | Assessed at baseline, immediately after baseline/post intervention, at two weeks, 2 months and 4 months.
  Assessed using the 14 item Hospital Anxiety and Depression Scale (HADS). HADS has an Anxiety subscale and a Depression subscale, each with 7 questions. Add the scores of each of the 7 questions of the Anxiety subscale for a total score on the Anxiety subscale. Add the scores of each of the 7 questions of the Depression subscale for a total score on the Depression subscale. Scores range, 0-21 on each subscale; score > 10 indicates clinical anxiety or depression; scores 8-10 indicate "borderline" anxiety or depression.
Acceptability | Assessed immediately after baseline/ post intervention, at two weeks, 2 months and 4 months.
  Assessed using a modified version of the an acceptability questionnaire developed by the Ottawa decision aid framework. Acceptability refers to ratings regarding the comprehensibility of components of a decision aid, its length, amount of information, balance in presentation of information about options, and overall suitability for decision making. Response options to individual items are poor, fair, good excellent, with good and excellent indicating a higher level of acceptability. This is not a scales responses can are reported descriptively for each item separately in terms of proportions responding positively or negatively on each criteria.
Time | Assessed at immediately after baseline/ post intervention, 2 months and 4 months.
  Measure of total time with Genetic counselor.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Bombard, PhD, Principal Investigator — St. Michael's Hospital and University of Toronto
Locations (3):
- Canada (3):
  - Sunnybrook Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to research who are interested in / conducting similar research in this field. This data will be available upon request, keeping with research ethics procedures.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: for 5 years after study has been completed and the trail data has been published.
Access Criteria: Data will be made available to research who are interested in / conducting similar research in this field. This data will be available upon request, keeping with research ethics procedures.
URL: http://stmichaelshospitalresearch.ca/labs/yvonne-bombard/

REFERENCES:
- [Derived] Shickh S, Hirjikaka D, Clausen M, Kodida R, Mighton C, Reble E, Sam J, Panchal S, Aronson M, Graham T, Armel SR, Glogowski E, Elser C, Eisen A, Carroll JC, Shuman C, Seto E, Baxter NN, Scheer A, Shastri-Estrada S, Feldman G, Thorpe KE, Schrader KA, Lerner-Ellis J, Kim RH, Faghfoury H, Bombard Y. Genetics Adviser: a protocol for a mixed-methods randomised controlled trial evaluating a digital platform for genetics service delivery. BMJ Open. 2022 Apr 29;12(4):e060899. doi: 10.1136/bmjopen-2022-060899. PMID 35487723